CLINICAL TRIAL: NCT03506815
Title: A Pilot Study Assessing the Feasibility of a Randomized Controlled Trial Investigating Primary Thromboprophylaxis With Rivaroxaban in Patients With Malignancy and Central Venous Catheters
Brief Title: Thromboprophylaxis With Rivaroxaban In Patients With Malignancy and Central Venous Lines
Acronym: TRIM-Line
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Queen Elizabeth II Health Sciences Centre (Other); University of Alberta (Other); Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 001
Record Dates: First submitted 2018-03-19; First posted 2018-04-24 (Actual); Results first posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2023-01

CONDITIONS: Upper Extremity Deep Vein Thrombosis; Central Venous Catheter Thrombosis; Cancer
Keywords: Upper Extremity Deep Vein Thrombosis; Thromboprophylaxis; Cancer; Randomized Trial
MeSH Terms: conditions — Upper Extremity Deep Vein Thrombosis; Neoplasms | interventions — Rivaroxaban

STUDY DESIGN:
Intervention Model Description: Randomized Pilot Trial comparing two groups - Rivaroxaban 10mg po daily for 90 days vs standard of care (usual treatment)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rivaroxaban Thromboprophylaxis (Experimental): Rivaroxaban 10 mg po daily for 90 days(+/- 3 days). After the Day - 90 follow up, the study treatment will be discontinued and subsequent treatment will be at the discretion of the attending physician.
  Interventions: Drug: Rivaroxaban 10 MG
- Standard of care (No Intervention): No rivaroxaban prophylaxis. Management will be at the discretion of the attending physician.

INTERVENTIONS:
Drug: Rivaroxaban 10 MG — Rivaroxaban 10mg po daily x 90 (+/- 3 days)
  Other Names: Xarelto 10mg tablet po daily
  Arms: Rivaroxaban Thromboprophylaxis

SUMMARY:
Purpose of the Pilot Trial:

To determine the feasibility of conducting a multicentre randomized open label controlled trial evaluating the use of prophylactic dose rivaroxaban to prevent central venous catheter (CVC) associated venous thromboembolism (VTE) among cancer patients.

Hypothesis: treatment with low dose rivaroxaban (10mg) will reduce the incidence of upper extremity venous thrombosis in a high risk population with cancer and CVC.

DETAILED DESCRIPTION:
Design:

This is a pilot interventional study to be conducted at 2 Canadian Centres. The Ottawa Hospital and Juravinski Hospital. It is an open label randomized controlled trial.

Consenting participants, meeting eligibility criteria will be randomized at the time of enrollment to one of two groups.

Rivaroxaban 10mg by mouth daily x 90 (+/- 3) days OR Standard of Care

Participants in the treatment arm will have study drug dispensed at Day 1 and take medication for 90 days or until CVC is removed. Follow up visits (in person or phone) will occur at Day 30 (+/- 3 days) and Day 90 (+/- 3 days). Overall, participants will be followed for 3 months. Adverse events will be collected for the first 90 days.

Outcomes The primary feasibility outcome for the pilot study is the number of participants recruited per centre per month. We will obtain baseline details of the patient's type, location and treatment of cancer, comorbidities and medications. Secondary feasibility outcomes of the pilot study will include, consent rates, loss to follow up, adherence to therapy defining 80% or greater medication taken as having good adherence to study drug, proportion of screened patients who meet eligibility criteria.

ELIGIBILITY:
Inclusion Criteria:

1.Patients 18 years of age or older with a new or existing diagnosis of cancer with a CVC inserted within the last 72 hours.

Exclusion Criteria:

1. CVC in place for >72 hours
2. Patient requires anticoagulation for other indication
3. Concomitant use of dual antiplatelet therapy
4. Prior VTE
5. Major bleeding event in the last 6 weeks
6. Patient on concomitant medication with known interaction with rivaroxaban (eg. CYP3A4 inhibitor)
7. Pregnancy (documentation of use of effective contraception if sexually active or negative B-Hcg required)
8. Known renal failure, based on Creatinine clearance <30 mL/min (Cockcroft-Gault) (in the previous 3 months)
9. Documented severe liver disease (eg. acute clinical hepatitis, chronic active hepatitis, cirrhosis or ALT >3ULN) ( in the previous 3 months)
10. Known thrombocytopenia < 50x 109/L (in the previous 3 months)
11. Allergy to rivaroxaban
12. Life expectancy <6 months
13. History of condition at increased bleeding risk including, but not limited to:

    1. Major surgical procedure or trauma within 30 days before the randomization visit
    2. Clinically significant gastrointestinal bleeding within 6 months before the randomization visit
    3. History of intracranial, intraocular, spinal, or atraumatic intra-articular bleeding
    4. Chronic hemorrhagic disorder
    5. Known intracranial neoplasm, arteriovenous malformation, or aneurysm
    6. Sustained uncontrolled hypertension: systolic blood pressure ≥180 mmHg or diastolic blood pressure ≥100 mmHg
14. Primary malignancy diagnosis of basal cell or squamous cell carcinoma of the skin or acute leukemia or myelodysplastic syndrome
15. Geographic inaccessibility
16. Refused or unable to obtain consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2020-05-14 (Actual); Study Completion 2020-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rick T Ikesaka, MD, Principal Investigator — Ottawa Hospital Research Institute / Division of Hematology- The Ottawa Hospital
Locations (1):
- The Ottawa Hospital General Campus, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Pilot Feasibility Study- no current plan to share individual participant data

REFERENCES:
- [Result] Ikesaka R, Siegal D, Mallick R, Wang TF, Witham D, Webb C, Carrier M; Canadian Venous Thromboembolism Research Network (CanVECTOR). Thromboprophylaxis with rivaroxaban in patients with malignancy and central venous lines (TRIM-Line): A two-center open-label pilot randomized controlled trial. Res Pract Thromb Haemost. 2021 May 5;5(4):e12517. doi: 10.1002/rth2.12517. eCollection 2021 May. PMID 34027291

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rivaroxaban Thromboprophylaxis | Standard of Care
Started | 52 | 53
Completed | 37 | 53
Not Completed | 15 | 0
Not completed — Adverse Event | 8 | 0
Not completed — End of chemotherapy removal of peripherally inserted central venous catheter | 5 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Elective Surgery | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rivaroxaban Thromboprophylaxis | Standard of Care | Total
Number analyzed (Participants) | 52 | 53 | 105
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (11.9) | 61.6 (12.7) | 60.8 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 36 | 72
  Male | 16 | 17 | 33
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 50 | 49 | 99
  Black | 0 | 1 | 1
  Asian | 0 | 3 | 3
  Other | 2 | 0 | 2
Cancer type [Count of Participants; unit: Participants]
  Breast | 15 | 14 | 29
  Colorectal | 15 | 16 | 31
  Stomach | 5 | 2 | 7
  Gynecological | 6 | 5 | 11
  Pancreas | 3 | 7 | 10
  Other | 8 | 9 | 17
Central Venous Catheter Type [Count of Participants; unit: Participants]
  PICC | 40 | 42 | 82
  Port-a-Cath | 12 | 11 | 23
Metastatic disease [Count of Participants; unit: Participants] | 14 | 19 | 33

OUTCOME MEASURES:

1. Primary Outcome: Primary Feasibility Outcome - Number of Participants Recruited Per Month
Description: A convenience sample size of 100 patients was chosen to allow reporting of the average monthly recruitment.
Time Frame: 12 months
Population: Total number of participants enrolled per site over a 12 month recruitment period.
Measure: Number; unit: Average enrolment rate/month/site
Groups:
- Site 1: Ottawa Hospital
- Site 2: Juravinski Hospital
Arm/Group | Site 1 | Site 2
Number analyzed (Participants) | 90 | 15
Average enrolment rate/month/site | 7.5 | 2.0

2. Secondary Outcome: Secondary Feasibility Outcomes - Percentage of Participants With Good Adherence to Therapy
Description: Good adherence defined as 80% or greater study medication taken in patients randomized to receive Rivaroxaban thromboprophylaxis.
Time Frame: 90 days
Population: Data not collected for participants in the "Standard of Care" arm since they did not receive study medication and management was left to the discretion of the attending physician.
Measure: Number; unit: percentage of participants
Arm/Group | Rivaroxaban Thromboprophylaxis | Standard of Care
Number analyzed (Participants) | 52 | 0
percentage of participants | 96.7 |

3. Other Pre Specified Outcome: Number of Participants With Thrombotic Complication
Description: Thrombotic complication was defined as a combination of major venous thromboembolism (VTE); any symptomatic or incidentally detected proximal deep vein thrombosis (DVT) of the lower or upper limbs, any nonfatal symptomatic or incidental pulmonary embolism (PE), and pulmonary embolism-related death) and any other deep (ie, distal, splanchnic, or cerebral) or superficial venous thrombosis.
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Rivaroxaban Thromboprophylaxis | Standard of Care
Number analyzed (Participants) | 52 | 53
Participants
  Major VTE | 2 | 3
  Major VTE - Upper extremity | 2 | 2
  Major VTE - PE | 0 | 1
  Other thrombotic event - splanchnic vein thrombosis | 1 | 1
  Other thrombotic event - superficial vein thrombosis | 0 | 1

4. Other Pre Specified Outcome: Number of Participants With CVC-Related Complication
Description: Central venous catheter (CVC) occlusion was defined as an obstruction of the CVC lumen that prevents or limits the ability to flush, withdraw blood, and/or administer solutions or medications
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Rivaroxaban Thromboprophylaxis | Standard of Care
Number analyzed (Participants) | 52 | 53
Participants
  CVC-associated infection | 0 | 2
  CVC migration | 0 | 1
  CVC positional occlusion | 0 | 1
  CVC occlusion | 0 | 1

5. Other Pre Specified Outcome: Number of Participants With Major Bleeding
Description: Defined by the International Society on Thrombosis and Haemostasis (ISTH) as overt bleeding associated with a decrease in the hemoglobin level of ≥2 g/dL, which led to transfusion of two or more units of packed red blood cells, occurred in a critical site, or contributed to death.
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Rivaroxaban Thromboprophylaxis | Standard of Care
Number analyzed (Participants) | 52 | 53
Participants | 1 | 0

6. Other Pre Specified Outcome: Number of Participants With Clinically Relevant Non-Major Bleed
Description: Clinically relevant non-major bleeding, as per the standardized definition by the ISTH, is any signs or symptoms of hemorrhage not meeting criteria for major bleeding but associated with medical intervention, unscheduled in-person contact with a healthcare professional or need for hospitalization or increased level of care.
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Rivaroxaban Thromboprophylaxis | Standard of Care
Number analyzed (Participants) | 52 | 53
Participants | 2 | 2

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Rivaroxaban Thromboprophylaxis | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/53
Serious Adverse Events (participants affected / at risk) | 11/52 | 10/53
Other Adverse Events (participants affected / at risk) | 16/52 | 12/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Rivaroxaban Thromboprophylaxis (N=52) | Standard of Care (N=53)
Major Bleed (Gastrointestinal disorders) | 1 (1) | 0 (0) — Participant with metastatic esophageal cancer (liver, bone, brain and lymph node metastases) had a Gastrointestinal Bleed leading to hospital admission and transfusion of 3 units of red blood cells.
Febrile Neutropenia (Blood and lymphatic system disorders) | 1/1 (1) | 0 (0) — Febrile Neutropenia
Fever (Immune system disorders) | 3 (3) | 0 (0) — Fever
Small Bowel Obstruction (Gastrointestinal disorders) | 3 (3) | 0 (0) — Small bowel obstruction
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) — Shortness of breath
Chest Pain (General disorders) | 0 (0) | 1 (1) — Chest Pain
Decreased O2 (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Decreased O2 saturation, req. O2, Query PE
Ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Diabetic Ulcer- Left foot
E-Coli, Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1) — E-Coli, Urinary Tract Infection
Pnemonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) — Fungal Pnemonia- Rivaroxaban arm Pnemonia- Standard of Care Recurrent Pnemonia- Standard of care
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) — Nausea & vomiting
Neutropenia Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1) — Neutropenia Enterocolitis
Renal Failure (Renal and urinary disorders) | 0 (0) | 1 (1) — Renal failure
Respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Upper Respitory Tract Infection
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rivaroxaban Thromboprophylaxis (N=52) | Standard of Care (N=53)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) — Anemia 1 case asymptomatic anemia
Common Cold (General disorders) | 1 (1) | 0 (0) — Common Cold
Chemotherapy Infusion Reaction (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) — Chemotherapy infusion reaction
Chest pain (General disorders) | 1 (1) | 1 (1) — Chest pain
Dizziness (General disorders) | 0 (0) | 1 (1) — Dizziness
Fever (General disorders) | 2 (2) | 1 (1) — Fever
GERD (Gastrointestinal disorders) | 0 (0) | 1 (1) — GERD
Herpes (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Herpes simplex vulva
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1) — Hydronephrosis
Indigestion (Gastrointestinal disorders) | 2 (2) | 0 (0) — Indigestion
Yeast Infection (Infections and infestations) | 0 (0) | 1 (1) — Intermittant yeast infections
Lower back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Lower back pain
Migraine (Nervous system disorders) | 1 (1) | 0 (0) — Migraine Headache
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Neck pain
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1) — Atrial Fibrillation
Radiation toxicity (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Radiation toxicity
Prolongation post chemo pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Prolongation post chemo pain
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) — adhesive rash =2 bilateral lower leg=1
Symptomatic Anemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) — Symptomatic Anemia
Syncope (General disorders) | 0 (0) | 1 (1) — Syncopal Episode
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (7) | 2 (3) — Thrombocytopenia
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 1 (1) — Urinary Tract Infection
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) — Urosepsis

LIMITATIONS AND CAVEATS:
A PROBE design was chosen in order to be pragmatic and to reflect standard clinical practice, which could make the results more easily applicable to routine medical care. The study was designed to assess feasibility and not to determine differences in the risk of clinical events between treatment groups. As a result, the number of clinical outcome events was relatively small, leading to imprecision and wide confidence intervals.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2019-09-18): https://cdn.clinicaltrials.gov/large-docs/15/NCT03506815/Prot_000.pdf